CLINICAL TRIAL: NCT04104776
Title: A Phase 1/2 Study of DZR123 (CPI-0209) in Patients With Advanced Solid Tumors and Lymphomas
Brief Title: A Study of Tulmimetostat DZR123 (CPI-0209) in Patients With Advanced Solid Tumors and Lymphomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDZR123A02101; CPI-0209-01 (Other: Constellation Pharmaceuticals); 2023-508002-20-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor; Diffuse Large B Cell Lymphoma; Lymphoma, T-Cell; Mesothelioma, Malignant; Prostatic Neoplasms, Castration-Resistant; Endometrial Cancer; Ovarian Clear Cell Carcinoma; Metastatic Castration-resistant Prostate Cancer
Keywords: Tulmimetostat; DZR123; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-cell; Lymphoma, T-cell; Lymphoma, Non-Hodgkin; Lymphoma; Neoplasms by Site; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Topoisomerase Inhibitors; Molecular Mechanisms of Pharmacological Action; Antineoplastic Agents; Endometrial Cancer; Ovarian Clear Cell Carcinoma; Food effect; Adenine-thymine (AT)-rich interactive domain-containing protein 1A (ARID1A); ARID1A wildtype (ARID1A WT) endometrial carcinoma; Metastatic castration-resistant prostate cancer (mCRPC)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell; Mesothelioma, Malignant; Prostatic Neoplasms, Castration-Resistant; Endometrial Neoplasms; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma; Neoplasms by Site; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Phase 1 (Experimental): Tulmimetostat will be dosed once per day orally in patients with advanced tumors.
  Interventions: Drug: Tulmimetostat
- Phase 2 Cohort M1 (Experimental): Tulmimetostat will be dosed once per day orally in 28 day cycles.
  • Cohort M1: patients with urothelial carcinoma or other advanced/metastatic solid tumors (with known ARID1A mutation)
  Interventions: Drug: Tulmimetostat
- Phase 2 Cohort M2 (Experimental): Tulmimetostat will be dosed once per day orally in 28 day cycles.
  • Cohort M2 patients with ovarian clear cell carcinoma (with known ARID1A mutation)
  Interventions: Drug: Tulmimetostat
- Phase 2 Cohort M3 (Experimental): Tulmimetostat will be dosed once per day orally in 28 day cycles.
  • Cohort M3 patients with endometrial carcinoma (with known ARID1A mutation)
  Interventions: Drug: Tulmimetostat
- Phase 2 Cohort M4 (Experimental): Tulmimetostat will be dosed once per day orally in 28 day cycles.
  • Cohort M4 patients with peripheral T-cell lymphoma (PTCL) and patients with diffuse large B-cell lymphoma (DLBCL), including patients with documented germinal center B cell like diffuse large B-cell lymphoma (GCB-DLBCL) with at least 1 Enhancer of Zeste Homolog 2 (EZH2) hotspot mutation
  Interventions: Drug: Tulmimetostat
- Phase 2 Cohort M5 (Experimental): Tulmimetostat will be dosed once per day orally in 28 day cycles.
  • Cohort M5 patients with relapsed or refractory malignant pleural or peritoneal mesothelioma with known BAP1 loss
  Interventions: Drug: Tulmimetostat
- Phase 2 Cohort M6 (Experimental): Tulmimetostat will be dosed once per day orally in 28 day cycles.
  • Cohort M6 patients with castration-resistant prostate cancer (mCRPC) with measurable soft tissue disease
  Interventions: Drug: Tulmimetostat
- Phase 2 Cohort M7 (Experimental): Tulmimetostat will be dosed once per day orally in 28 day cycles.
  • Cohort M7 food effect in patients with ARID1A wildtype (ARID1A WT) endometrial carcinoma
  Interventions: Drug: Tulmimetostat
- Phase 1 Cohort M8 (Experimental): Tulmimetostat will be dosed once per day orally in combination with enzalutamide Cohort M8 patients with castration-resistant prostate cancer (mCRPC).
  Interventions: Drug: Tulmimetostat
- Phase 2 Cohort M8 (Experimental): Tulmimetostat will be dosed once per day orally in 28-day cycles in combination with enzalutamide.
  • Cohort M8 patients with castration-resistant prostate cancer (mCRPC).
  Interventions: Drug: Tulmimetostat; Drug: Enzalutamide

INTERVENTIONS:
Drug: Tulmimetostat — Tulmimetostat dosed once per day orally in 28 day cycles
  Other Names: DZR123
Drug: Enzalutamide — Enzalutamide dosed once per day orally in 28 day cycles
  Arms: Phase 2 Cohort M8

SUMMARY:
The purpose of this open-label, first-in-human (FIH) trial is to evaluate the safety, tolerability, and preliminary clinical activity of Tulmimetostat as a monotherapy in patients with advanced solid tumors and lymphomas.

DETAILED DESCRIPTION:
The study is divided into Phase 1 and Phase 2. In Phase 1 and the Phase 2 expansion (M1 to M7), patients are non-randomized. In Phase 2 optimization, patients in Cohort M2 and M3 (Stage 2a and 2b) and Cohort M8 (Part 2) are randomized.

Phase 1 of the study is composed of a Tulmimetostat Dose Escalation period in patients with advanced tumors and aims to determine maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of Tulmimetostat as monotherapy in patients with advanced tumors.

Phase 2 of the study is planned to evaluate safety and tolerability and antitumor activity of Tulmimetostat in six disease-specific cohorts (M1 to M6). Patients in Cohorts M1, M2, M3, M5, and M6 will be enrolled at 10 to 29 patients per cohort, using a Simon 2-stage design. Cohort M4 will enroll up to 20 patients with lymphoma in a single-stage.

The primary aim of Phase 2 part of the study is to evaluate the antitumor activity of Tulmimetostat, and characterize the safety and tolerability of Tulmimetostat as monotherapy in patients with selected tumors.

In Phase 2, two additional doses are planned to be evaluated in cohorts M2 and M3 in 2 stages: Stage 2a and Stage 2b. In Stage 2a approximately 20 patients will be enrolled per cohort and will be randomized 1:1 to receive 2 prespecified dose levels of Tulmimetostat once daily. When protocol criteria for initiating Stage 2b will be fulfilled after completion of Stage 2a, then Stage 2b will be opened for enrolment of additional 10 patients in one or both dose arms in each of the two cohorts. Thus, up to 40 patients per cohort (M2 and M3) could be enrolled.

The study will explore the Tulmimetostat in anti-tumor activity and effect of food on pharmacokinetics of Tulmimetostat in in patients with ARID1A WT endometrial carcinoma (Cohort M7) and safety and anti-tumor activity of Tulmimetostat in in combination with enzalutamide in patients with mCRPC (Cohort M8).

In Cohort M8 Part 1, the safety and tolerability of Tulmimetostat in and enzalutamide combination will be evaluated in patients with mCRPC. The M8 Part 1 dose escalation incorporates combination of Tulmimetostat in at escalating provisional doses with enzalutamide.

In Cohort M8 Part 2, the safety, tolerability and preliminary antitumor activity of Tulmimetostat at a RP2D in combination with enzalutamide will be further evaluated in patients with mCRPC.

ELIGIBILITY:
Key Inclusion Criteria:

* Eligible Phase 1 patients are adults who have a confirmed locally advanced or metastatic tumors (solid tumors or lymphoma) that have relapsed following standard therapy or progressed through standard therapy or who have a disease for which no standard effective therapy exists.
* Eligible Phase 2 patients in cohorts M1 to M3 are adults who are known to have the ARID1A mutation by next-generation sequencing (NGS) testing; have measurable disease per Response Evaluation Criteria in Solid Tumors 1.1 and who have confirmed relapsed urothelial or other advanced/metastatic solid tumors (M1), ovarian clear cell carcinoma (M2), or endometrial carcinoma (M3).
* Eligible Phase 2 patients in Cohort M4 are adults who have either relapsed or refractory PTCL (at least 10 patients) or DLBCL (up to 10 patients), including patients with documented GCB DLBCL with EZH2 hotspot mutation. Patients with PTCL must have at least 1 prior line of therapy and patients with DLBCL must have at least 2 prior lines of standard therapy; and are not considered candidates to receive CAR-T or ASCT therapy.
* Eligible Phase 2 patients in Cohort M5 are adults who are known to the have the BAP1 loss, have malignant pleural or peritoneal mesothelioma, and have progressed on at least 1 prior line of active therapy.
* Eligible Phase 2 patients in Cohort M6 are adults who have mCRPC with measurable soft tissue disease with CT scan as defined by PCWG3 criteria, have baseline testosterone levels ≤ 50 ng/dL (≤ 2.0 nM) and have surgical or ongoing medical castration and who have progressed on at least 1 androgen-receptor signaling inhibitor and at least 1 taxane-based chemotherapy (cabazitaxel, France only).
* Eligible Phase 2 patients in Cohort M7 are adults with recurrent, advanced ARID1A WT endometrial carcinoma confirmed by NGS testing and have measurable disease per Response Evaluation Criteria in Solid Tumors 1.1 Patients will be enrolled with maximum up to 2 prior lines of systemic therapy for treating endometrial carcinoma that must include at least one treatment line with systemic platinum-based chemotherapy in advanced/ recurrent disease setting, and anti-programmed cell death protein 1 (PD-1)/ anti-programmed death-ligand 1 (PD-L1) therapy, either in combination or separately, unless these are contraindicated or are not locally accessible.
* Eligible Part 1 and Part 2 patients in Cohort M8 are adults who have mCRPC with measurable soft tissue disease as per PCWG3 criteria, have baseline testosterone levels ≤ 50 ng/dL (≤ 2.0 nM), have surgical or ongoing medical castration or hormone sensitive prostate cancer (HSPC) disease stage. In addition, Eligible part 1 patients in Cohort M8 may have received abiraterone treatment in mCRPC while eligible part 2 patients in Cohort M8 must have received abiraterone treatment in mCRPC. In addition, only for M8 Part 1: Patients may have received no more than one previous regimen of taxane-based chemotherapy in mCRPC or HSPC setting. For M8 Part 2: Patients may have received no more than one previous regimen of taxane-based chemotherapy in HSPC setting. Patients for both M8 Part 1 and M8 Part 2 must have evidence of prostate cancer progression (per PCWG3) and must have ongoing ADT (androgen deprivation therapy) with a GnRH analogue, antagonist or bilateral orchiectomy (i.e., surgical or medical castration).
* All patients will have Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 and adequate organ function.

Key Exclusion Criteria:

1. Medical Conditions

   * Previous solid organ or allogeneic hematopoietic cell transplantation (HCT).
   * Known symptomatic untreated brain metastases. Patients with central nervous system (CNS) metastases must have stable neurologic status following local therapy for at least 4 weeks on a stable or decreasing dose of steroids (≤ 10 mg daily prednisone or equivalent). Patients in the M4 lymphoma cohort are excluded if they have known CNS involvement by lymphoma.
   * Clinically significant cardiovascular disease, including:

     * Myocardial infarction or stroke within 3 months (6 months for M8 cohort) prior to Day 1 of treatment.
     * Unstable angina within 3 months (6 months for M8 cohort) prior to Day 1 of treatment.
     * Congestive heart failure or cardiomyopathy with New York Heart Association (NYHA) Class 3 or 4.
     * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes).
     * Uncontrolled hypertension despite 2 concomitant antihypertensive therapies.
     * For Cohorts M1-M6: QT interval corrected by the Fridericia correction formula (QTcF) > 480 msec on the Screening ECG.
     * For Cohorts M7 and M8: QTcF interval ≥ 450 msec at screening.
   * Major surgery within 4 weeks before starting study drug or not recovered from any effects of prior major surgery (uncomplicated central line placement or fine needle aspirate are not considered major surgery).
   * Gastrointestinal disorders that may significantly interfere with the absorption of the study medication, such as ulcerative colitis, malabsorption syndrome, refractory nausea and vomiting, biliary shunt, significant bowel resection.
   * Uncontrolled active infection requiring intravenous antibiotic, antiviral, or antifungal medications within 14 days before the first dose of study drug. Controlled infections on concurrent antimicrobial agents and antimicrobial prophylaxis per institutional guidelines are acceptable.
   * Suspected pneumonitis or interstitial lung disease (confirmed by radiography or CT) or a history of these conditions.
   * History of a concurrent or second malignancy except for certain adequately treated cancers such as local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease, adequately treated Stage 1 or 2 cancer currently in complete remission, or any other cancer in complete remission for ≥ 3 years. Patients with a history of T-cell lymphoblastic lymphoma or T-cell lymphoblastic leukemia are not eligible.
   * Current known active or chronic infection with HIV, hepatitis B, or hepatitis C. Screening for these viruses is not required unless there is a past history or current suspicion of viral hepatitis.
   * Clinically active or symptomatic viral hepatitis or chronic liver disease.
   * Unstable or severe uncontrolled medical condition or any important medical or psychiatric illness or abnormal laboratory finding that would increase the risk to the patient associated with participation in the study.
   * For Cohort M7 Only: Patients not willing to or cannot remain fasted due to a medical condition for 2 hours before and 1 hour after dose administration.
2. Prior/Concomitant Therapy:

   * Prior Anticancer Treatment:

     * Systemic Anticancer Treatment: Patients must not have received chemotherapy, targeted therapy, small molecules, antibodies, investigational anticancer therapy, or other anticancer therapeutics (except gonadotropin-releasing hormone analogues) within 4 weeks (or 5 half-lives, whichever is shorter) before the first dose of the study drug. For nitrosoureas or mitomycin C, a 6-week washout is required. For prior PD-1 or PD-L1 therapy, a washout period of at least 4 weeks is acceptable. All toxicities from prior therapies must have resolved to Grade 1 or less, except for endocrinopathies requiring medication, neuropathy, and alopecia, which must have resolved to Grade 2 or less.
     * EZH2 Inhibitor: Previous treatment with an EZH2 inhibitor is not allowed.
     * Radiation Therapy: Patients must not have received radiation therapy (including radiofrequency ablation) within 4 weeks before the first dose of the study drug. However, a single fraction of radiotherapy for palliation confined to one field is permitted within 1 week prior to Day 1 of treatment.
     * Stereotactic Body Radiation Therapy: Patients must not have received this therapy within 2 weeks before the first dose of the study drug.
     * Chemoembolization or Radioembolization: Patients must not have received these treatments within 4 weeks before the first dose of the study drug.
   * Concomitant Medication:

     * CYP3A4/5 Inducers or Inhibitors: Patients must not take strong CYP3A4/5 inducers or inhibitors (except enzalutamide in Cohort M8) within 7 days or 5 times the reported half-life of the CYP3A4/5 inhibitor or inducer (whichever is longer) prior to the first dose of the study drug and for the duration of the study.
3. Other Exclusions

   * General Exclusions:

     * Pregnancy and Breastfeeding: Patients who are breastfeeding, pregnant (as confirmed by a serum β-hCG pregnancy test within 72 hours prior to the first dose of the study drug), or planning to conceive or father children during the trial and for 183 days after the last dose of the study drug are excluded. Women of nonchildbearing potential (post-menopausal for more than 1 year or surgically sterilized) do not require a serum pregnancy test. A highly sensitive urine test can be used if a serum test is not appropriate. Female patients with false-positive β-hCG values may be enrolled with written consent from the Sponsor's Medical Monitor after pregnancy has been excluded.
     * Compliance: Patients who are unwilling or unable to comply with the study protocol or requirements are excluded.
   * Additional Exclusions for Cohort M6 (mCRPC) Only:

     * Bone-only Disease: Patients with bone-only disease without nodal disease and no evidence of visceral spread are excluded.
     * Structurally Unstable Bone Lesions: Patients with bone lesions that are structurally unstable and concerning for impending fracture are excluded.
     * Herbal Products: Patients using herbal products that may decrease prostate-specific antigen (PSA) levels within 4 weeks prior to Day 1 of treatment and during the study are excluded.
     * Prostate Cancer Treatments: Patients who have received the following treatments for prostate cancer within the specified timeframes prior to Day 1 of treatment are excluded:

       1. First-generation androgen receptor antagonists (e.g., bicalutamide, nilutamide, flutamide) within 4 weeks.
       2. 5α reductase inhibitors, ketoconazole, estrogens (including diethylstilbestrol), or progesterones within 2 weeks.
     * Planned Palliative Procedures: Patients with planned palliative procedures for alleviation of bone pain, such as radiation therapy or surgery, are excluded.
4. Additional Exclusion Criteria for Cohort M8 (DZR123 and Enzalutamide Combination in mCRPC) only:

   * Biochemical recurrence/prostate-specific antigen (PSA)-only disease.
   * Prior Enzalutamide Treatment:

     * For M8 Part 1: Patients who have received prior enzalutamide.
     * For M8 Part 2: Patients who have received prior enzalutamide, apalutamide, darolutamide, or any other investigational androgen receptor pathway inhibitor (ARPi).
   * Herbal Products: Use of herbal products that may decrease PSA levels within 4 weeks prior to Day 1 of treatment and during the study.
   * Planned Palliative Procedures: Planned palliative procedures for alleviation of bone pain, such as radiation therapy or surgery.
   * Investigational Agents: Treatment with any investigational agent within 4 weeks before Day 1 of M8 Part 1 or M8 Part 2.
   * Bone Marrow Irradiation: Prior irradiation to more than 25% of the bone marrow.
   * Gastrointestinal Conditions: Active inflammatory gastrointestinal disease, chronic diarrhea, known diverticular disease, or previous gastric resection or lap band surgery. Gastroesophageal reflux disease under treatment with proton pump inhibitors is allowed.
   * Seizure History: History of seizure, loss of consciousness, or transient ischemic attack within 12 months of study entry, or any condition that may predispose to seizure (e.g., stroke, brain arteriovenous malformation, head trauma, underlying brain injury).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2030-02-27 (Estimated); Study Completion 2030-02-27 (Estimated)

PRIMARY OUTCOMES:
Tulmimetostat Monotherapy Phase 1: Frequency of Dose-limiting toxicities (DLTs) | DLTs assessed during Cycle 1 (cycle = 28 days)
  The maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of Tulmimetostat as monotherapy in patients with advanced tumors.
Tulmimetostat Monotherapy Phase 2: Overall response rate (ORR) | Up to 30 months
  ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) based on RECIST 1.1 or applicable response criteria
Cohort M8 Part 1: Frequency of Dose-limiting toxicities (DLTs) | DLTs assessed during Cycle 1 (cycle = 28 days)
  The maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of Tulmimetostat in combination with enzalutamide in patients with castration-resistant prostate cancer (mCRPC) with measurable soft tissue disease.
Cohort M8 Part 2: Overall response rate (ORR) | Up to 30 months
  ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) per Investigator assessment based on Prostate Cancer Clinical Trials Working Group 3 (PCWG3)

SECONDARY OUTCOMES:
Tulmimetostat Monotherapy Phase 1: Incidence Rate of AEs | Up to 18 months
  Number of Participants With Adverse Events (AEs)
Tulmimetostat Monotherapy Phase 1: Maximum observed plasma concentration (Cmax) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 1: Time of maximum observed plasma concentration (Tmax) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 1: Area under the plasma concentration-time curve from time zero to the last quantifiable time point (AUC0-last) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 1: Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-Inf) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 1: Terminal elimination half-life (T1/2) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 1: Plasma concentrations prior to the next dose-trough (Cmin) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 1: Gene expression in blood cells | Up to 18 months
  To characterize the Pharmacodynamics (PD) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 1: H3K27me3 | Up to 18 months
  To characterize the Pharmacodynamics (PD) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 1: Objective Response Rate (ORR) | Up to 30 months
  ORR defined as proportion of patients with a best overall response of complete response (CR) or partial response (PR), per Investigator assessment based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1 or applicable response criteria)
Tulmimetostat Monotherapy Phase 1: ORR per Gynecologic Cancer Intergroup (GCIG) | Up to 30 months
  ORR per Gynecologic Cancer Intergroup (GCIG)-defined CA-125 response criteria (ovarian cancer patients)
Tulmimetostat Monotherapy Phase 1: ORR per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) | Up to 30 months
  ORR per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) (in Phase 1 prostate cancer patients only)
Tulmimetostat Monotherapy Phase 1: Progression-free survival (PFS) | Up to 30 months
  PFS defined as the time from first dose to confirmed disease progression or death
Tulmimetostat Monotherapy Phase 1: Duration of response (DOR) | Up to 30 months
  DOR defined as the time from the date of first response to the date of confirmed disease progression
Tulmimetostat Monotherapy Phase 1: Time to response (TTR) | Up to 30 months
  TTR defined as the time from first dose to date of first response
Tulmimetostat Monotherapy Phase 1: Disease Control Rate (DCR) | Up to 30 months
  DCR defined as the proportion of patients with a best overall response of CR, PR, or stable disease (SD)
Tulmimetostat Monotherapy Phase 2: Progression-free survival (PFS) | Up to 30 months
  PFS defined as the time from first dose to confirmed disease progression or death
Tulmimetostat Monotherapy Phase 2: Time-to-progression (TTP) | Up to 30 months
  TTP defined as duration from the start of treatment until the disease progression
Tulmimetostat Monotherapy Phase 2: Duration of response (DOR) | Up to 30 months
  DOR defined as the time from the date of first response to the date of confirmed disease progression
Tulmimetostat Monotherapy Phase 2: Time to response (TTR) | Up to 30 months
  TTR defined as the time from first dose to date of first response
Tulmimetostat Monotherapy Phase 2: Disease Control Rate (DCR) | Up to 30 months
  DCR defined as the proportion of patients with a best overall response of CR, PR, or SD per cohort and Tulmimetostat dose level
Tulmimetostat Monotherapy Phase 2: ORR per Gynecologic Cancer Intergroup (GCIG) | Up to 30 months
  ORR per GCIG-defined CA-125 response criteria (ovarian cancer patients)
Tulmimetostat Monotherapy Phase 2: Overall survival (OS) | Up to 30 months
  OS defined as the time from first dose to death
Tulmimetostat Monotherapy Phase 2: Incidence Rate of AEs | Up to 18 months
  Number of Participants With Adverse Events (AEs)
Tulmimetostat Monotherapy Phase 2: Maximum observed plasma concentration (Cmax) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 2: Time of maximum observed plasma concentration (Tmax) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 2: Area under the plasma concentration-time curve from time zero to the last quantifiable time point (AUC0-last) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 2: Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-Inf) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 2: Terminal elimination half-life (T1/2) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 2: Plasma concentrations prior to the next dose-trough (Cmin) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 2: Gene expression in blood cells | Up to 18 months
  To further characterize the Pharmacodynamics (PD) profile of Tulmimetostat as monotherapy
Tulmimetostat Monotherapy Phase 2: H3K27me3 | Up to 18 months
  To further characterize the Pharmacodynamics (PD) profile of Tulmimetostat as monotherapy
Cohort M7: Maximum observed plasma concentration (Cmax) | Up to 18 months
  To evaluate the effect of a High-fat high-calorie (HFHC) meal on the Pharmacokinetic (PK) behavior of Tulmimetostat monotherapy dose in patients with ARID1A WT endometrial carcinoma
Cohort M7: Time of maximum observed plasma concentration (Tmax) | Up to 18 months
  To evaluate the effect of a High-fat high-calorie (HFHC) meal on the Pharmacokinetic (PK) behavior of Tulmimetostat monotherapy dose in patients with ARID1A WT endometrial carcinoma
Cohort M7: Area under the plasma concentration-time curve from time zero to the last quantifiable time point (AUC0-last) | Up to 18 months
  To evaluate the effect of a High-fat high-calorie (HFHC) meal on the Pharmacokinetic (PK) behavior of Tulmimetostat monotherapy dose in patients with ARID1A WT endometrial carcinoma
Cohort M7: Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-Inf) | Up to 18 months
  To evaluate the effect of a High-fat high-calorie (HFHC) meal on the Pharmacokinetic (PK) behavior of Tulmimetostat monotherapy dose in patients with ARID1A WT endometrial carcinoma
Cohort M7: Terminal elimination half-life (T1/2) | Up to 18 months
  To evaluate the effect of a High-fat high-calorie (HFHC) meal on the Pharmacokinetic (PK) behavior of Tulmimetostat monotherapy dose in patients with ARID1A WT endometrial carcinoma
Cohort M7: Plasma concentrations prior to the next dose-trough (Cmin) | Up to 18 months
  To evaluate the effect of a High-fat high-calorie (HFHC) meal on the Pharmacokinetic (PK) behavior of Tulmimetostat monotherapy dose in patients with ARID1A WT endometrial carcinoma
Cohort M8 Part 1: Incidence Rate of AEs | Up to 18 months
  Number of Participants With Adverse Events (AEs)
Cohort M8 Part 1: Maximum observed plasma concentration (Cmax) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 1: Time of maximum observed plasma concentration (Tmax) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 1: Area under the plasma concentration-time curve from time zero to the last quantifiable time point (AUC0-last) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 1: Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-Inf) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 1: Plasma concentrations prior to the next dose-trough (Cmin) | Up to 18 months
  To characterize the Pharmacokinetic (PK) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 1: Gene expression in blood cells | Up to 18 months
  To characterize the Pharmacodynamics (PD) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 1: H3K27me3 | Up to 18 months
  To characterize the Pharmacodynamics (PD) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 1: Objective Response Rate (ORR) | Up to 30 months
  ORR defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) per Investigator assessment based on Prostate Cancer Clinical Trials Working Group 3 (PCWG3)
Cohort M8 Part 1: Duration of response (DOR) | Up to 30 months
  DOR defined as the time from the date of first response to the date of disease progression per PCWG3.
Cohort M8 Part 1: Disease Control Rate (DCR) | Up to 30 months
  DCR defined as the proportion of patients with a best overall response of CR, PR, or stable disease (SD) per PCWG3.
Cohort M8 Part 1: Prostate-Specific Antigen 50 (PSA50) Response | Up to 18 months
  PSA50 response defined as PSA decline by >=50% from baseline
Cohort M8 Part 1: Number of participants experiencing Dose-limiting toxicities (DLTs) | DLTs assessed during Cycle 1 (cycle = 28 days)
  To establish dose-toxicity relationship between Tulmimetostat and enzalutamide combination
Cohort M8 Part 2: Incidence Rate of AEs | Up to 18 months
  Number of Participants With Adverse Events (AEs)
Cohort M8 Part 2: Maximum observed plasma concentration (Cmax) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 2: Time of maximum observed plasma concentration (Tmax) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 2: Area under the plasma concentration-time curve from time zero to the last quantifiable time point (AUC0-last) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 2: Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-Inf) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 2: Plasma concentrations prior to the next dose-trough (Cmin) | Up to 18 months
  To further characterize the Pharmacokinetic (PK) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 2: Gene expression in blood cells | Up to 18 months
  To further characterize the Pharmacodynamics (PD) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 2: H3K27me3 | Up to 18 months
  To further characterize the Pharmacodynamics (PD) profile of Tulmimetostat and enzalutamide
Cohort M8 Part 2: Duration of response (DOR) | Up to 30 months
  DOR defined as the time from the date of first response to the date of confirmed disease progression.
Cohort M8 Part 2: Progression-free survival (PFS) | Up to 30 months
  PFS assessed by PCWG3, and defined as the time from first dose to confirmed disease progression or death
Cohort M8 Part 2: Prostate-Specific Antigen 50 (PSA50) Response | Up to 18 months
  PSA50 response defined as PSA decline by >=50% from baseline
Cohort M8 Part 2: Time to Prostate-Specific Antigen (PSA) Progression | Up to 18 months
  Time to PSA progression defined as the time from first dose to PSA progression
Cohort M8 Part 2: Overall survival (OS) | Up to 30 months
  OS defined as the time from first dose to death in patients with mCRPC

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (60):
- United States (17):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Maryland - Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - South Texas Accelerated Research Therapeutics (Start) - Midwest Location, Grand Rapids, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Langone Medical Center - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer, Seattle, Washington
- France (8):
  - Bergonie Institute, Bordeaux
  - Oscar Lambret Center, Lille
  - Leon Berard Center, Lyon
  - Nantes University Hospital Center - Hotel Dieu Hospital (Satellite), Nantes
  - Nantes University Hospital Center - Hotel Dieu Hospital, Nantes
  - Nord Laennec Hospital, Saint-Herblain
  - Strasbourg Europe Institut of Cancerology, Strasbourg
  - Gustave Roussy, Villejuif
- Italy (5):
  - Irccs University Hospital of Bologna, Bologna
  - National Cancer Institute, IRCCS, Milan
  - European Institute of Oncology (IEO), IRCCS, Milan
  - University Polyclinic Foundation "Agostino Gemelli" - IRCCS, Rome
  - Gruppo Humanitas - Humanitas Research Hospital - Cancer Center, Rozzano
- Poland (5):
  - University Teaching Centre, Early Clinical Trials Unit, Gdansk
  - Polish Mother's Memorial Hospital-Research Institute, Lodz
  - University Teaching Hospital in Poznan, Department of Gynecologic Oncology, Poznan
  - Medical Center Pratia Poznan, Skorzewo
  - Maria Sklodowska-Curie - National Research Institute of Oncology, Warsaw
- South Korea (7):
  - Keimyung University - Dongsan Medical Center, Daegu
  - National Cancer Center, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
- Spain (11):
  - University Hospital Vall d'Hebron, Barcelona
  - University Hospital of Girona Dr. Josep Trueta, Girona
  - University Clinic of Navarra - Madrid, Madrid
  - University Hospital 12 de Octubre, Madrid
  - University Hospital Quiron Madrid, Madrid
  - University Hospital Son Espases, Palma de Mallorca
  - University Clinic of Navarra - Pamplona, Pamplona
  - University Clinical Hospital of Salamanca, Salamanca
  - University Hospital Complex of Santiago (CHUS), Santiago de Compostela
  - University Hospital Virgen del Rocio (HUVR), Seville
  - Valencia Oncology Institute (IVO), Valencia
- United Kingdom (7):
  - Royal United Hospital, Bath
  - University Hospitals of Leicester NHS Trust, Leicester
  - Royal Marsden Hospital - London, London
  - Imperial College Healthcare NHS Trust, London
  - The Christie NHS Foundation Trust, Department of Medical Oncology, Manchester
  - Royal Marsden Hospital - Sutton, Sutton
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com